CLINICAL TRIAL: NCT06689670
Title: To Evaluate the Safety and Performance of INT001 in the Percutaneous Ablation of Liver Tumors: A Prospective, Single-arm, Single-center Clinical Study
Brief Title: Needle-based Percutaneous Ablation of Liver Tumors.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: inTumo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: inTumoThera
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Liver Tumors; HCC - Hepatocellular Carcinoma; Metastatic Liver Tumor
Keywords: liver; tumor; ablation; needle; out-patient
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Arm, Open-label, Single-Center Clinical Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INT001 Treatment (Experimental): Patients with liver tumors enrolled in the study will receive INT001
  Interventions: Device: Needle based delivery of INT001 into liver tumors under real-time image guidance

INTERVENTIONS:
Device: Needle based delivery of INT001 into liver tumors under real-time image guidance — Using ultrasound or CT imaging, the liver tumor is located. Under local anesthesia or, if necessary, intravenous sedation, the needle is inserted through the skin and the needle tip is brought to the center of the liver tumor using image guidance. 1-2 ml of the INT-001 is injected. The needle is removed and a bandaid is applied to the skin entry site. Right after, or as soon as MRI becomes available, MRI is performed to show that the entire tumor has been treated.
  Other Names: Percutaneous tumor ablation

SUMMARY:
The goal of this clinical trial is to learn if INT001 can ablate liver tumors in adults in an outpatient setting. It will also help us learn about the safety of INT001. The main questions it aims to answer are:

1. Using a needle under image guidance, the liver tumor is accessed and INT001 is injected. Upon injection into tumor, does INT001 ablate/kill the tumor entirely?
2. What medical problems do participants experience when receiving INT001?

Participants will:

Receive INT001 on day 1. Visit the clinic day 7, 30 and 90. Receive lab tests during each visit and MRI on day 30 and 90.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary or secondary liver cancer.
2. ECOG Performance Status score of 0 - 2
3. Age ≥18 years, <100 years
4. Life expectancy of ≥3 months
5. Patient is unsuitable for surgical resection or transplantation
6. Ability of the patient to understand and sign the Informed Consent Form describing the study's nature
7. Volunteer's willingness and ability to comply with protocol requirements, including all procedures, clinical evaluations, and follow-up visits

Exclusion Criteria:

1. Decompensated liver function, specifically Child-Pugh C, moderate to severe ascites, coagulopathy, or severe cirrhosis.
2. Signs of liver dysfunction: AST or ALT >5 times the upper limit of normal (ULN), Serum bilirubin level >2.0 mg/dL
3. Individuals with bleeding disorders.
4. History of allergy or intolerance to contrast agents to be used during imaging for assessing treatment efficacy after INT001 application.
5. Patients with life-threatening serious extrahepatic disease.
6. Patients with concurrent conditions that, in the investigator's opinion, would prevent clinical benefit from the study procedure or could compromise patient safety or study objectives (including but not limited to ongoing infection, renal dysfunction, or morbidity).
7. Significant medical or psychiatric illness.
8. Pregnant or breastfeeding women or women planning to conceive within the next 6 months.
9. Patients participating in another study investigating a device, drug, or procedure that may impact the study treatment outcome.
10. Lesions that do not show contrast uptake on contrast-enhanced CT or MR angiography.
11. Lesions that are not hypervascular on angiography.
12. Patients who do not have CT or MR imaging available at the screening visit or are unwilling or unable to undergo MRI for various reasons during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ablation | MRI will be performed the day of the intervention, at 30 days and at 90 days.
  Ablation of the tumor will be assessed using imaging criteria such as RECIST.
Adverse events | From day 1 to day 90
  Procedure-Related and Post-Procedure Complications Complications related to the procedure and the postoperative period

SECONDARY OUTCOMES:
Biomarkers | Day 30 and Day 90
  Biomarkers such as AFP will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Selcukbiricik, MD, Principal Investigator — Koc University Hospital
Locations (1):
- Koc University Hospital, Topkapı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Keum H, Albadawi H, Zhang Z, Graf E, Santos PRD, Gunduz S, Oklu R. Bioengineered Ionic Liquid for Catheter-Directed Tissue Ablation, Drug Delivery, and Embolization. Adv Mater. 2024 Jun;36(23):e2309412. doi: 10.1002/adma.202309412. Epub 2024 Feb 16. PMID 38305472
- [Result] Cevik E, Albadawi H, Zhang Z, Demirlenk Y, Atar D, Keum C, Kim J, Graf E, Gunduz S, Rehman S, Oklu R. Catheter-Directed Ionic Liquid Embolic Agent for Rapid Portal Vein Embolization, Segmentectomy, and Bile Duct Ablation. Adv Mater. 2024 Jul;36(29):e2402570. doi: 10.1002/adma.202402570. Epub 2024 May 7. PMID 38678378
- [Result] Demirlenk YM, Albadawi H, Zhang Z, Atar D, Cevik E, Keum H, Kim J, Rehman S, Gunduz S, Graf E, Mayer JL, Dos Santos PR, Oklu R. Prostate tissue ablation and drug delivery by an image-guided injectable ionic liquid in ex vivo and in vivo models. Sci Transl Med. 2024 Jul 3;16(754):eadn7982. doi: 10.1126/scitranslmed.adn7982. Epub 2024 Jul 3. PMID 38959326
- [Result] Albadawi H, Zhang Z, Keum H, Cevik E, Nagalo BM, Gunduz S, Kita H, Oklu R. Percutaneous Delivery of Oncogel for Targeted Liver Tumor Ablation and Controlled Release of Therapeutics. Adv Mater. 2024 Nov;36(45):e2406080. doi: 10.1002/adma.202406080. Epub 2024 Aug 15. PMID 39148179